CLINICAL TRIAL: NCT04161118
Title: Phase II Trial of TisaGenlecleucel in Elderly Patients With First-Relapsed or Primary Refractory Aggressive B-cell Non-Hodgkin Lymphoma
Brief Title: TisaGenlecleucel in Elderly Patients With First-Relapsed or Primary Refractory Aggressive B-cell Non-Hodgkin Lymphoma
Acronym: TIGER-CTL019
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of the funding agreement by the financial sponsor of the study. Small number of patients enrolled, none of the planned analyses will be feasible to draw conclusions on the safety or efficacy of the therapy.
Sponsor: University of Cologne (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Trial Chairman, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-3903
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (CTL019) (Experimental): All patients will receive a single target dose of 0.6 to 6.0 × 108 of autologous tisagenlecleucel (CTL019) transduced T-cells with a viability of at least 70% administered via IV infusion after optional bridging with chemo- or immunotherapy and lymphodepleting (LD) chemotherapy with cyclophosphamide and fludarabine.
  Interventions: Drug: CTL019

INTERVENTIONS:
Drug: CTL019 — IV Infusion

SUMMARY:
A phase II trial of TisaGenlecleucel (CTL019) in Elderly Patients with First-Relapsed or Primary Refractory Aggressive B-cell Non-Hodgkin Lymphoma

DETAILED DESCRIPTION:
This is a single-arm, prospective, multicenter phase-II trial for elderly patients with aNHL failing 1st-line treatment with immunochemotherapy containing rituximab and anthracycline, who are not eligible for either autologous or allogeneic stem cell transplantation, defined as age > 65 years, or > 60 years old with HCT-CI score >2. This trial evaluates the CMR rate 12 weeks after tisagenlecleucel (CTL019) infusion, the incidence and severity of adverse events, progression-free survival, and overall survival after one and two years after tisagenlecleucel (CTL019).

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed and dated informed consent must be obtained prior to participation in the study
2. Patients with first relapse of aggressive B-cell Non-Hodgkin Lymphoma (aNHL) within 365 days after rituximab- and anthracycline-containing first-line immunochemotherapy or aNHL refractory to first-line therapy (not achieving a CR or PR), who are ineligible for either autologous or allogeneic stem cell transplantation, defined by age > 65 years, or > 60 years with a HCT-CI score > 2 (https://qxmd.com/calculate/calculator_108/hematopoietic-cell-transplantation-specific-comorbidity-index-hct-ci) and not older than 80 years.
3. Histologically confirmed (by local histopathological assessment) aNHL at relapse or progression due to refractory disease after front line therapy. aNHL is defined by the following list of subtypes:

   1. DLBCL, NOS (GCB, ABC, centroblastic, immunoblastic, anaplastic)
   2. FL grade 3B
   3. T-cell-rich/histiocyte-rich large B-cell lymphoma (T/HRBCL)
   4. DLBCL associated with chronic inflammation
   5. Intravascular large B-cell lymphoma
   6. ALK+ large B-cell lymphoma
   7. B-cell lymphoma, unclassifiable, (with features intermediate between DLBCL and classical HL)
   8. High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
   9. High-grade B-cell lymphoma, NOS
   10. HHV8+ DLBCL, NOS
   11. DLBCL transformed from follicular lymphoma
   12. DLBCL transformed from marginal zone lymphoma
   13. DLBCL, leg type
4. Measurable disease:

   1. Nodal lesions >15 mm in the long axis, regardless of the length of the short axis, and/or
   2. Extranodal lesions (outside lymph node or nodal mass, but including liver and spleen) >10 mm in long AND short axis
5. ECOG performance status 0-2
6. Adequate organ function:

   a. Kidney function defined as: i. Serum creatinine estimated glomerular filtration rate GFR ≥ 30mL/min b. Hepatic function defined as: i. ALT and AST ≤ 5 × ULN, except for aNHL-related functional impairment. ii. Bilirubin ≤2.0 mg/dl except for patients with Gilbert syndrome, who may be included if their total bilirubin is ≤3.0 × ULN and direct bilirubin ≤1.5 × ULN OR for aNHL-related functional impairment c. Adequate bone marrow function (regardless of transfusion) defined as: i. WBC ≥2500/µL ii. Absolute neutrophil count (ANC) >1000/µL iii. Platelets ≥50,000/µL iv. Hemoglobin >8.0 g/dl d. Minimum level of pulmonary function defined as: i. No or mild dyspnea (≤ Grade 1) ii. pulse oxygenation ≥ 91% on room air
7. Life expectancy of more than six months
8. Women have to be in menopausal or post-menopausal status or confirmed as not having potential on childbearing
9. Male participants with female partners of childbearing potential are eligible to participate if they agree to contraceptive methods as described in the study protocol

Exclusion Criteria:

1. Patients with Richter's transformation, Burkitt lymphoma, or primary CNS lymphoma (PCNSL)
2. Prior treatment with anti-CD19 therapy, adoptive T-cell therapy, or any prior gene therapy product
3. Treatment with any lymphoma-directed second-line anticancer therapy prior to enrollment with the exception of intermittent steroid therapy. After enrollment, bridging therapy is permitted for disease control.
4. Patients with active CNS involvement are excluded, except if the CNS involvement has been effectively treated (i.e. patient is asymptomatic) and local treatment was >4 weeks before enrollment
5. Prior allogeneic bone marrow transplantation (HSCT)
6. Active hepatitis B, hepatitis C, or hepatitis E infection
7. HIV-positive patients
8. Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
9. Any of the following cardiovascular conditions:

   1. Unstable angina, myocardial infarction, coronary artery bypass graft (CABG), or stroke within 6 months prior to screening,
   2. LVEF <45% as determined by ECHO at screening except for aNHL-related functional impairment,
   3. NYHA functional class III or IV (Chavey et al. 2001) at screening,
   4. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II) and third degree AV block, unless adequately controlled by pacemaker implantation,
   5. Resting QTcF ≥450 msec (male) or ≥460 msec (female) at screening or inability to determine the QTcF interval,
   6. Risk factors for Torsades de Point (TdP), including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia, or any of the following:
   7. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or
   8. Concomitant medication(s) with a "Known Risk of Torsades de Point" per www.qtdrugs.org that cannot be discontinued or replaced by safe alternative medication.
10. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
    2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
    3. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    4. Adequately treated carcinoma in situ without evidence of of recurrence for at least 3 years prior to the study
    5. A primary malignancy which has been completely resected and in complete remission for ≥ 3 years
11. Pregnant or nursing (lactating) women and women who are not confirmed to be menopausal/post-menopausal. Or women who are capable of giving birth.
12. Intolerance to the excipients of the tisagenlecleucel cell product
13. Active or history of inflammatory disorders or autoimmune disease that required systemic steroids or immunosuppressive medications, with exception of vitiligo or resolved childhood asthma
14. Active tuberculosis
15. Exposure to any investigational agent(s) within 4 weeks prior to study entry
16. Chemotherapy less than 2 weeks before leukapheresis
17. Simultaneous radiotherapy to tisagenlecleucel infusion (radiotherapy between leukapheresis and day -6 before tisagenlecleucel infusion is permitted)
18. Ongoing necessity for systemic corticosteroids >10mg daily prednisone equivalent. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
19. History of active primary immunodeficiency
20. Major surgery (defined as opening at least one body cavity) within 4 weeks prior to study entry
21. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening CT scan
22. Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PDL2, anti-CTLA-4 antibodies, other immune checkpoint inhibitors
23. Prior treatment with any anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy.
24. Current treatment within another therapeutic clinical trial with experimental and not approved drugs and treatment combinations
25. Patient's lack of accountability and inability to appreciate the nature, meaning and consequences of the trial and to formulate his/her own wishes correspondingly
26. Non-compliance, e.g. due to

    1. Drug dependency or substance abuse that would interfere with cooperation with requirements of the trial
    2. Refusal of blood products during treatment
    3. Change of residence to abroad
    4. any similar circumstances that appear to make protocol treatment or long-term follow-up impossible
27. Patients who have a relationship of dependence or employer-employee relationship to the sponsor or the investigator
28. Committal to an institution on judicial or official order

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Estimation of the efficacy of treatment with tisagenlecleucel (CTL019) in elderly patients with r/r aNHL by measuring the complete metabolic response (CMR) rate 12 weeks after tisagenlecleucel (CTL019) infusion | 12 weeks after tisagenlecleucel (CTL019) infusion
  Estimation of the efficacy of treatment with tisagenlecleucel (CTL019) in elderly patients with r/r aNHL by measuring the complete metabolic response (CMR) rate 12 weeks after tisagenlecleucel (CTL019) infusion

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From study start to study end (44 months)
  Incidence and severity of adverse events (AEs)
Progression-free survival (PFS) rates at 1 and 2 year(s) | Up to two years from study start
  Progression-free survival (PFS) rates at 1 and 2 year(s)
Overall survival (OS) rates at 1 and 2 year(s) | Up to two years from study start
  Overall survival (OS) rates at 1 and 2 year(s)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University of Cologne, Cologne
  - Universitätsklinik Essen, Klinik für Hämatologie, Essen

IPD SHARING:
Plan to Share IPD: No